CLINICAL TRIAL: NCT02055820
Title: A Phase Ib/II, Open-Label Study Evaluating the Safety, Efficacy and Pharmacokinetics of GDC-0199 (ABT-199) in Combination With Rituximab (R) or Obinutuzumab (G) Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) in Patients With B-Cell Non-Hodgkin's Lymphoma (NHL) and DLBCL
Brief Title: A Study Evaluating the Safety, Efficacy and Pharmacokinetics of Venetoclax Combined With Chemotherapy in Participants With B-Cell Non-Hodgkin's Lymphoma (NHL) and DLBCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO27878; 2013-003749-40 (EudraCT Number)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — venetoclax; Cyclophosphamide; obinutuzumab; Rituximab; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venetoclax + G-CHOP Arm (Experimental): Phase I: Participants will receive 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle will consist of 21 days. Phase II: Participants will receive 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + obinutuzumab. Each cycle will consist of 21 days. For both phase I and II, participants with ongoing response without excessive toxicity may receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
  Interventions: Drug: Venetoclax; Drug: Cyclophosphamide; Drug: Obinutuzumab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Venetoclax + R-CHOP Arm (Experimental): Phase I: Participants will receive 6 cycles of CHOP and 8 cycles of venetoclax + rituximab. Each cycle will consist of 21 days. Phase II: Participants will receive 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + rituximab. Each cycle will consist of 21 days. For both phase I and II, participants with ongoing response without excessive toxicity may receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
  Interventions: Drug: Venetoclax; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Venetoclax — Venetoclax 200 to 800 milligrams (mg) tablets will be administered orally once daily (QD) on Days 4-10 of Cycle 1 and Days 1-10 of Cycles 2-8 during Phase I and MTD will be administered according to the same schedule during Phase II.
  Other Names: GDC-0199, ABT-199
Drug: Cyclophosphamide — Cyclophosphamide 750 milligrams per square meter (mg/m^2) administered intravenously (IV) on Day 1 of each 21-day cycle up to Cycle 6.
Drug: Obinutuzumab — Obinutuzumab will be administered by IV infusion as an absolute dose of 1000 mg on Days 1, 8, 15 of Cycle 1 and Day 1 of Cycles 2-8 (cycle length = 21 days).
  Arms: Venetoclax + G-CHOP Arm
Drug: Rituximab — Rituximab 375 mg/m^2 dose will be administered IV on Day 1 of every 21-day cycle.
  Other Names: MabThera/Rituxan
  Arms: Venetoclax + R-CHOP Arm
Drug: Doxorubicin — Doxorubicin 50 mg/m^2 administered IV on Day 1 of each 21-day cycle up to Cycle 6.
Drug: Vincristine — Vincristine 1.4 mg/m^2 (maximum 2 mg) administered IV on Day 1 of each 21-day cycle up to Cycle 6.
Drug: Prednisone — Prednisone 100 mg per day orally on Days 1-5 of each 21-day cycle up to Cycle 6.

SUMMARY:
This is a multicenter, open-label, dose-finding study of venetoclax administered orally in combination with rituximab (R) or obinutuzumab (G) and standard doses of cyclophosphamide, doxorubicin, vincristine and oral prednisone (CHOP) in participants with Non-Hodgkin's Lymphoma (NHL). The study consisted of 2 stages: a dose-finding Phase Ib stage and a Phase II expansion stage. In the Phase I portion of the study, participants were randomized to one of 2 treatment arms venetoclax in combination with R-CHOP (Arm A) and venetoclax in combination with G-CHOP (Arm B) and explored the doses of venetoclax in combination with R-CHOP and G-CHOP. The maximum tolerated dose (MTD) of venetoclax in combination with R-CHOP and G-CHOP was determined during the dose-finding stage. For the Phase II portion of the study, the venetoclax dose for venetoclax + R-CHOP was on a non-continuous dosing schedule as determined by the Phase Ib portion of the study based on safety and tolerability observed in participants treated in the dose escalation portion of the study. On 17 July 2016, Roche/Genentech as the sponsor of Study BO21005 (Goya study), a Phase III study that evaluated G CHOP versus R-CHOP in 1L DLBCL, informed through a press release that the primary endpoint of investigator-assessed PFS was not met. Given these results, Arm B (venetoclax + G-CHOP) was not expanded in Phase II in patients who are first-line with DLBCL.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* At least one bi-dimensionally measurable lymphoma lesion on CT scan defined as > 1.5 cm in its longest dimension, which is also FDG avid by screening PET scan.
* Confirmed availability of archival or freshly biopsied tumor tissue prior to study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate hematologic function
* For female participants of childbearing potential, agreement to use highly effective forms of contraception

Dose-Escalation Portion of the Study:

* Participants must have histologically confirmed B-cell NHL, except MCL or SLL
* Participants must have never received previous R-CHOP treatment
* Any relapsed/refractory participants that are enrolled during the dose escalation should have received only a single previous treatment regimen

Expansion Portion of the Study:

* Participants must have previously untreated CD20-positive DLBCL and IPI score must be 2-5

Exclusion Criteria:

General Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to receive any of the individual components of CHOP, rituximab or obinutuzumab
* Prior anthracycline therapy
* Participants with ongoing corticosteroid use >30 mg per day of prednisone or equivalent
* CNS lymphoma or primary mediastinal DLBCL
* Vaccination with live vaccines within 28 days prior to randomization
* Chemotherapy or other investigational therapy within 28 days prior to the start of Cycle 1
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled concomitant disease
* Significant cardiovascular disease or significant pulmonary disease
* Left ventricular ejection fraction less than (<) 50% as defined by multiple-gated acquisition (MUGA)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1 Day 1
* Received the following agents within 7 days prior to the first dose of venetoclax: steroid therapy for anti-neoplastic intent; strong and moderate cytochrome P450 (CYP) 3A4 inhibitors or inducers; grapefruit/grapefruit products, seville oranges or star fruit within 3 days prior to the first dose of venetoclax
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Recent major surgery
* Women who are pregnant or lactating

Dose-Escalation Portion of the Study:

* Participants with confirmed mantle cell lymphoma (MCL) or small lymphocytic lymphoma (SLL)

Expansion Portion of the Study:

* Participants with transformed lymphoma (participants with discordant bone marrow involvement (i.e., low grade histology in bone marrow) may be considered after discussion with the Medical Monitor)
* Prior therapy for NHL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2013-11-17 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (52):
- United States (9):
  - St. Jude Heritage Healthcare, Fullerton, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Central Coast Medical Oncology, Santa Maria, California
  - The West Clinici, St Louis, Missouri
  - Hackensack University Medical Center; WFAN - Imus Pediatric Center, Hackensack, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Uni of Rochester Medical Center; Wilmot Cancer Center, Pharmacy Department, Rochester, New York
  - Tennessee Oncology, Nashville, Tennessee
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, CSI, Kelowna, British Columbia
  - BC Cancer Agency Vancouver Centre - PARENT; BC Cancer Agency, Vancouver, British Columbia
  - Jewish General Hospital; Research Unit, Montreal, Quebec
  - CHU de Quebec - Hôpital de l' Enfant Jésus, Québec
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Vseobecna Fakultni Nemocnice v Praze, I. Interni Klinika - Klinika Hematoonkologie VFN a 1. LF UK, Prague
- France (11):
  - Hopital Henri Mondor, Unite Hemopathies lymphoides, Créteil
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Clinique Victor Hugo; Pharmacie, Le Mans
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hopital Saint Eloi, Montpellier
  - CHU Nantes - Hôtel Dieu; Service Assistance Medicale à la Procreation, Nantes
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel; Hematologie, Rouen
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem; Belgyogyaszati Klinika Hematologiai Tanszek, Debrecen
- Italy (5):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliero Universitaria San Martino, Genoa, Liguria
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera Vincenzo Cervello, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Pisana; U.O. Farmaceutica, Pisa, Tuscany
- Netherlands (3):
  - Amsterdam UMC Location VUMC, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht, Utrecht
- Spain (6):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals; Hematology, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario de Salamanca, Salamanca

REFERENCES:
- [Result] Zelenetz AD, Salles G, Mason KD, Casulo C, Le Gouill S, Sehn LH, Tilly H, Cartron G, Chamuleau MED, Goy A, Tam CS, Lugtenburg PJ, Petrich AM, Sinha A, Samineni D, Herter S, Ingalla E, Szafer-Glusman E, Klein C, Sampath D, Kornacker M, Mobasher M, Morschhauser F. Venetoclax plus R- or G-CHOP in non-Hodgkin lymphoma: results from the CAVALLI phase 1b trial. Blood. 2019 May 2;133(18):1964-1976. doi: 10.1182/blood-2018-11-880526. Epub 2019 Mar 8. PMID 30850381
- [Derived] Samineni D, Huang W, Gibiansky L, Ding H, Zhang R, Li C, Sinha A, Rajwanshi R, Humphrey K, Bazeos A, Salem AH, Miles D. Population Pharmacokinetics and Exposure-Response Analyses for Venetoclax in Combination with R-CHOP in Relapsed/Refractory and Previously Untreated Patients with Diffuse Large B Cell Lymphoma. Adv Ther. 2022 Jan;39(1):598-618. doi: 10.1007/s12325-021-01919-z. Epub 2021 Nov 25. PMID 34822104
- [Derived] Morschhauser F, Feugier P, Flinn IW, Gasiorowski R, Greil R, Illes A, Johnson NA, Larouche JF, Lugtenburg PJ, Patti C, Salles GA, Trneny M, de Vos S, Mir F, Samineni D, Kim SY, Jiang Y, Punnoose E, Sinha A, Clark E, Spielewoy N, Humphrey K, Bazeos A, Zelenetz AD. A phase 2 study of venetoclax plus R-CHOP as first-line treatment for patients with diffuse large B-cell lymphoma. Blood. 2021 Feb 4;137(5):600-609. doi: 10.1182/blood.2020006578. PMID 33538797

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At start the trial had a randomised-controlled component, until July 2016 once the arm B (Gazyva) got closed following the publication of results of another trial. Since July 2016, the trial was single-arm, not randomised anymore, and kept including patients in only 1 arm (Arm A, rituximab).
Pre-assignment Details: The data reported for participant flow is based on safety population, which includes all participants who received at least one dose of study medication.
Groups:
- Venetoclax 200 mg +R-CHOP; Venetoclax 400 mg +R-CHOP; Venetoclax 600 mg +R-CHOP; Venetoclax 800 mg +R-CHOP: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + rituximab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 800 mg +R-CHOP Phase II: Phase II: Participants received 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + rituximab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 200 mg +G-CHOP; Venetoclax 400 mg +G-CHOP; Venetoclax 600 mg +G-CHOP: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 800 mg + G-CHOP A: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. In this arm venetoclax was administered as follows: Cycle 1 Days 4-10; Cycles 2-8 Days 1-10, Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 800 mg +G-CHOP B: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. In this arm venetoclax was administered as follows: Cycle 1 Days 4-8; Cycles 2-8 Days 1-5. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Period: Phase I: Dose-Finding
Arm/Group | Venetoclax 200 mg +R-CHOP | Venetoclax 400 mg +R-CHOP | Venetoclax 600 mg +R-CHOP | Venetoclax 800 mg +R-CHOP | Venetoclax 800 mg +R-CHOP Phase II | Venetoclax 200 mg +G-CHOP | Venetoclax 400 mg +G-CHOP | Venetoclax 600 mg +G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg +G-CHOP B
Started | 7 | 3 | 8 | 6 | 0 | 7 | 7 | 6 | 6 | 6
Completed | 6 | 3 | 7 | 3 | 0 | 5 | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Period: Phase II: Expansion
Arm/Group | Venetoclax 200 mg +R-CHOP | Venetoclax 400 mg +R-CHOP | Venetoclax 600 mg +R-CHOP | Venetoclax 800 mg +R-CHOP | Venetoclax 800 mg +R-CHOP Phase II | Venetoclax 200 mg +G-CHOP | Venetoclax 400 mg +G-CHOP | Venetoclax 600 mg +G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg +G-CHOP B
Started | 0 | 0 | 0 | 0 | 208 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 159 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 49 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 33 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venetoclax 200 mg +R-CHOP | Venetoclax 400 mg +R-CHOP | Venetoclax 600 mg +R-CHOP | Venetoclax 800 mg +R-CHOP | Venetoclax 800 mg +R-CHOP Phase II | Venetoclax 200 mg +G-CHOP | Venetoclax 400 mg +G-CHOP | Venetoclax 600 mg +G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg +G-CHOP B | Total
Number analyzed (Participants) | 7 | 3 | 8 | 6 | 208 | 7 | 7 | 6 | 6 | 6 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (9.2) | 61.0 (13.1) | 57.0 (9.5) | 56.3 (11.9) | 61.4 (12.8) | 52.1 (16.2) | 60.9 (6.3) | 66.7 (4.2) | 60.5 (13.7) | 66.8 (6.7) | 61.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 94 | 2 | 5 | 4 | 4 | 2 | 120
  Male | 4 | 1 | 6 | 4 | 114 | 5 | 2 | 2 | 2 | 4 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 6 | 1 | 2 | 3 | 151 | 6 | 3 | 4 | 5 | 6 | 187
  Unknown or Not Reported | 1 | 2 | 6 | 3 | 53 | 1 | 4 | 2 | 1 | 0 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 4
  White | 6 | 1 | 2 | 2 | 154 | 7 | 2 | 4 | 5 | 4 | 187
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 6 | 4 | 42 | 0 | 4 | 2 | 1 | 2 | 64

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs were reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0). Decrease in B cells, lymphopenia, and leukopenia caused by lymphopenia were not considered DLTs but instead were expected outcomes of study treatment. Any Grade >/= 3 adverse event, that was attributed to having a reasonable possibility of being related to the combined administration of venetoclax plus R-CHOP or G-CHOP, that could not be attributed by the investigator to an alternative, clearly identifiable cause such as tumor progression, concurrent illness or medical condition, or concomitant medication and that occurred during the DLT observation period (start of venetoclax treatment through end of Cycle 2) was considered a DLT for dose-escalation purposes. Grade 3 or 4 neutropenia or thrombocytopenia identified on Day 1 of Cycle 2 or 3, resulting in dose delay were considered DLTs.
Time Frame: Start of venetoclax administration (Cycle 1 Day 4 or 3 days after first CHOP dose) up to end of Cycle 2 (cycle length = 21 days)
Population: Safety population: All participants who enrolled in the study and received any amount of venetoclax or R-CHOP/G-CHOP were included in the safety population for safety analyses. Here, participants in the Dose Finding phase were analyzed.
Measure: Number; unit: Participants
Groups:
- Venetoclax 200 mg + R-CHOP; Venetoclax 400 mg + R-CHOP; Venetoclax 600 mg + R-CHOP; Venetoclax 800mg + R-CHOP: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + rituximab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 200mg + G-CHOP; Venetoclax 400mg + G-CHOP; Venetoclax 600mg + G-CHOP: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 800 mg + G-CHOP A: Venetoclax + G-CHOP 800 mg A Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. In this arm venetoclax was delivered in Cycle 1 on Days 4-10 and Cycles 2-8 on Days 1-10. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax 800 mg + G-CHOP B: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. In this arm ventoclax was delivered in Cycle 1 on Days 4-8 and Cycles 2-8 on Days 1-5. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg + G-CHOP B
Number analyzed (Participants) | 7 | 3 | 8 | 6 | 7 | 7 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0

2. Primary Outcome: Percentage of Previously Untreated DLBCL Participants With Complete Response (CR) Defined by Positron Emission Tomography-Computed Tomography (PET/CT) Scan Using the Modified Lugano Classification Assessed by Independent Review Committee (IRC)
Description: CR was defined as follows according to modified Lugano classification for PET/CT-based response: Lymph nodes and extra-lymphatic sites with score 1, 2, or 3 with or without a residual mass on 5-point scale with 1) no uptake above background; 2) uptake </= mediastinum; 3) uptake < mediastinum but </= liver. No evidence of fluorodeoxyglucose (FDG)-uptake disease in marrow. If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy
Time Frame: Baseline up to end of treatment (up to approximately 6 months)
Population: Intent-to-treat (ITT) population: All participants who enrolled in the study were included in the ITT population. Data reported for all participants for whom data were available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Venetoclax + R-CHOP 800 mg Phase II: Phase II: Participants received 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + rituximab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax + R-CHOP 800 mg Phase II
Number analyzed (Participants) | 211
Percentage of participants | 68.2 [61.50 to 74.47]

3. Primary Outcome: Percentage of Participants With CR Defined by PET/CT Scan in Previously Untreated DLBCL Co-Expressing Both Bcl-2 and c-Myc Proteins (DE-DLBCL) Participants Assessed by IRC
Description: as for outcome 2
Time Frame: Baseline up to end of treatment (up to approximately 6 months)
Population: Intent-to-treat (ITT) population: All participants who enrolled in the study were included in the ITT population. Data reported for subgroup of the ITT, DE Participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Venetoclax + R-CHOP 800 mg Phase II
Number analyzed (Participants) | 81
Percentage of participants | 66.7 [55.32 to 76.76]

4. Secondary Outcome: Venetoclax Plasma PK: Area Under the Plasma Concentration-Time Curve (AUC)
Description: AUC was calculated based on measurement of venetoclax concentration in plasma over time. Venetoclax exposure was pooled across Phase I and II for the R-CHOP 800 mg cohorts.
  Data are reported as hour*micrograms per milliliter (hr*mcg/mL)
Time Frame: Predose (within 30 minutes) & 2, 4, 6, 8 hours (Hr) postdose on Cycle 1 Day 4 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. Reporting according to study drug received. One participant mistakenly received only 100 mg instead of the planned 200 mg dose and was reported in a separate arm for PK outcome measures.
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Groups:
- Venetoclax + R-CHOP 800 mg: Phase I and II: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + rituximab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax + G-CHOP 800mg: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax 800mg + R-CHOP | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax + R-CHOP 800 mg | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax + G-CHOP 800mg
Number analyzed (Participants) | 1 | 6 | 4 | 8 | 124 | 7 | 7 | 6 | 10
hr*mcg/mL | .66 (NA) — N/A as there is only one participant in this cohort | 2.51 (.97) | 3.87 (2.41) | 3.70 (1.59) | 4.51 (2.32) | 2.55 (1.13) | 4.33 (1.31) | 5.13 (2.41) | 6.20 (1.71)

5. Secondary Outcome: Venetoclax Plasma PK: Time to Maximum Observed Plasma Concentration (Tmax)
Description: Tmax was determined based on measurement of venetoclax concentrations in plasma over time. Venetoclax exposure was pooled across Phase I and II for the R-CHOP 800 mg cohorts.
Time Frame: Predose (within 30 minutes) & 2, 4, 6, 8 Hr postdose on Cycle 1 Day 4 (cycle length = 21 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hour
Groups:
- Venetoclax + R-CHOP 100 mg; Venetoclax 200 mg + R-CHOP; Venetoclax 400 mg + R-CHOP; Venetoclax 600 mg + R-CHOP; Venetoclax 800mg + R-CHOP: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + rituximab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
- Venetoclax + G-CHOP 800 mg: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax + R-CHOP 100 mg | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax + G-CHOP 800 mg
Number analyzed (Participants) | 1 | 6 | 4 | 8 | 124 | 7 | 7 | 6 | 10
Hour | 4.0 (NA) — N/A as there is only one participant in this cohort | 4.59 (1.08) | 6.50 (1.91) | 5.52 (2.07) | 5.53 (1.55) | 5.72 (1.42) | 6.56 (1.51) | 5.30 (2.38) | 5.79 (1.47)

6. Secondary Outcome: Venetoclax Plasma PK: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax was determined based on measurement of venetoclax concentrations in plasma over time. Venetoclax exposure was pooled across Phase I and II for the R-CHOP 800 mg cohorts.
  Data are reported as micrograms per milliliter
Time Frame: Predose (within 30 minutes) & 2, 4, 6, 8 Hr postdose on Cycle 1 Day 4 (cycle length = 21 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ug/ML
Arm/Group | Venetoclax + R-CHOP 100 mg | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax + G-CHOP 800 mg
Number analyzed (Participants) | 1 | 6 | 4 | 8 | 124 | 7 | 7 | 6 | 10
Ug/ML | .09 (NA) — N/A as there is only one participant in this cohort | .58 (.32) | .92 (.64) | .85 (.33) | 1.15 (.48) | .52 (.21) | 1.26 (.30) | 1.00 (.58) | 1.54 (.37)

7. Secondary Outcome: Venetoclax Plasma PK: Minimum Plasma Concentration (Cmin) Within the Dosing Interval
Description: Cmin was determined based on measurement of venetoclax concentrations in plasma over time. Venetoclax exposure was pooled across Phase I and II for the R-CHOP 800 mg cohorts.
Time Frame: Predose (within 30 minutes) & 2, 4, 6, 8 Hr postdose on Cycle 1 Day 4 (cycle length = 21 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Venetoclax + R-CHOP 100 mg | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax + G-CHOP 800 mg
Number analyzed (Participants) | 1 | 3 | 2 | 4 | 126 | 7 | 5 | 5 | 6
mcg/mL | 0.0714 (0.00) | 0.522 (0.441) | 0.253 (0.247) | 0.387 (0.141) | 0.640 (0.451) | 0.134 (0.107) | 0.395 (0.381) | 0.612 (0.535) | 0.628 (0.395)

8. Secondary Outcome: Prednisone Plasma PK: AUC
Description: AUC was determined based on measurement of Predisone concentrations in plasma over time.
Time Frame: Predose (within 30 minutes) and 0.5, 1, 2, 4, 6 Hr after prednisone dose on Day 1 of Cycle 1 and 2 (cycle length = 21 days)
Population: PK evaluable population: All participants who received study drug and provided at least one post-treatment PK sample. A similar dose strength of prednisone (100 mg) was administered across the treatment arms/venetoclax dose groups. Hence, the data are presented as an overall summary in Cycles 1 and 2.
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Groups:
- Venetoclax PK Popluation: All participants in the study.
  Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. Phase II: Participants received 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + obinutuzumab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax PK Popluation
Number analyzed (Participants) | 54
hr*mcg/mL
  Cycle 1, Day 1: number analyzed (Participants) | 52
  Cycle 1, Day 1 | 195 (72.8)
  Cycle 2, Day 1 | 184 (81.2)

9. Secondary Outcome: Prednisone Plasma PK: Tmax
Description: Tmax was determined based on measurement of Predisone concentrations in plasma over time.
Time Frame: as for outcome 8
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. A similar dose strength of prednisone (100 mg) was administered across the treatment arms/venetoclax dose groups. Hence, the data are presented as an overall summary in Cycles 1 and 2.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Venetoclax PK Popluation
Number analyzed (Participants) | 54
Hour
  Cycle 1, Day 1: number analyzed (Participants) | 52
  Cycle 1, Day 1 | 2.19 (1.61)
  Cycle 2, Day 1 | 3.80 (2.52)

10. Secondary Outcome: Prednisone Plasma PK: Cmax
Description: Cmax was determined based on measurement of Predisone concentrations in plasma over time.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Ng/ML
Arm/Group | Venetoclax PK Popluation
Number analyzed (Participants) | 54
Ng/ML
  Cycle 1, Day 1: number analyzed (Participants) | 52
  Cycle 1, Day 1 | 49.9 (28.7)
  Cycle 2, Day 1 | 43.2 (17.6)

11. Secondary Outcome: Rituximab PK: Cmax
Description: Cmax was determined using the post-dose rituximab plasma concentrations at the 800 mg Venetoclax Dose using the end of infusion time point on Cycle 1 Day 1.
Time Frame: End of Infusion on Cycle 1 Day 1 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. The Cmax of rituximab is presented at the 800 mg Venetoclax dose group. Hence, the data is not presented by the treatment arms/Venetoclax dose groups.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Venetoclax 800 mg: All participants in the study, who received 800 mg venetoclax.
  Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days. Phase II: Participants received 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + obinutuzumab. Each cycle consisted of 21 days. Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax 800 mg
Number analyzed (Participants) | 7
mcg/mL | 173 (39.4)

12. Secondary Outcome: Rituximab PK: Cmin Within the Dosing Interval
Description: Cmin was determined using the pre-dose rituximab plasma concentrations at the 800 mg Venetoclax Dose on Day 1 of Cycle 2.
Time Frame: Pre-dose on Cycle 2 Day 1 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. The Cmin of rituximab is presented at the 800 mg Venetoclax dose group. Hence, the data is not presented by the treatment arms/Venetoclax dose groups.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Venetoclax 800 mg
Number analyzed (Participants) | 8
mcg/mL | 26.1 (13)

13. Secondary Outcome: Obinutuzumab PK: Cmax
Description: Cmax was determined using the post-dose obinutuzumab plasma concentrations at the 800 mg Venetoclax Dose using the end of infusion time point on Cycle 1 Day 1.
Time Frame: End of Infusion on Cycle 1 Day 1 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. The Cmax of obinutuzumab is presented at the 800 mg Venetoclax dose group. Hence, the data is not presented by the treatment arms/Venetoclax dose groups.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Venetoclax 800 mg
Number analyzed (Participants) | 10
mcg/mL | 326 (76)

14. Secondary Outcome: Cyclophosphamide PK: Cmax
Description: Cmax was determined using the post-dose Cyclophosphamide plasma concentrations on Cycle 1 Day 1.
Time Frame: End of Infusion on Cycle 1 Day 1 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. Given a single dose strength of Cyclophosphamide was administered across the different Venetoclax dose groups and treatment arms, hence the data are presented as an overall summary.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Venetoclax PK Popluation
Number analyzed (Participants) | 36
mcg/mL | 32.1 (7.51)

15. Secondary Outcome: Doxorubicin PK: Cmax
Description: Cmax was determined using the post-dose Doxorubicin plasma concentrations.
Time Frame: End of Infusion on Cycle 1 Day 1 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. Given a single dose strength of Doxorubicin was administered across the different Venetoclax dose groups and treatment arms, hence the data are presented as an overall summary.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Venetoclax PK Popluation
Number analyzed (Participants) | 24
mcg/mL | 1260 (911)

16. Secondary Outcome: Vincristine PK: Cmax
Description: Cmax was determined using the post-dose Vincristine plasma concentrations.
Time Frame: End of Infusion on Cycle 1 Day 1 (cycle length = 21 days)
Population: PK evaluable population: All patients who received study drug and provided at least one post-treatment PK sample for whom data were available. Given a single dose strength of Vincristine was administered across the different Venetoclax dose groups and treatment arms, hence the data are presented as an overall summary.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Venetoclax PK Popluation
Number analyzed (Participants) | 28
mcg/mL | 54.0 (44.6)

17. Secondary Outcome: Percentage of Participants With Objective Response Defined as Partial Response (PR) or Complete Response (CR) Defined by Positron Emission Tomography-Computed Tomography (PET/CT) Using the Modified Lugano Classification Assessed by IRC
Description: Objective Response defined as PR (partial response) or CR (complete response) at end of treatment.
  CR: Lymph nodes and extra-lymphatic sites with score 1, 2 or 3 on a 5-point scale (with a higher score being a worse outcome). No evidence of fluorodeoxyglucose (FDG)-uptake disease in marrow. If the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
  PR: Lymph nodes and extralymphatic sites with score of 4 or 5 on the 5-point scale with reduced uptake compared with baseline and residual mass(es) of any size. CT-based response criteria for PR must also be met. No new lesions. In bone marrow residual uptake could be higher than in normal marrow but must be reduced compared with baseline; persistent focal changes in the marrow to be considered for further evaluation with magnetic resonance imaging (MRI) or biopsy or an interval scan. OR=PR+CR
Time Frame: Baseline to end of treatment (up to approximately 6 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Venetoclax + R-CHOP 800 mg Phase II
Number analyzed (Participants) | 211
Percentage of Participants | 81.5 [75.61 to 86.51]

18. Secondary Outcome: Percentage of Participants Who Are Alive and Without Disease Progression at Month 12
Description: Progressive disease (PD) was determined using the modified Lugano classification criteria. For PET-CT-based PD: Score 4 (uptake moderately > liver) or 5 (uptake markedly higher than liver and/or new lesions) with an increase in intensity of uptake from baseline in target nodes and nodal lesions, new FDG-uptake foci of extranodal lesions consistent with lymphoma at interim or end-of-treatment assessment, no non-measured lesions, new FDG-uptake foci consistent with lymphoma, new or recurrent FDG-uptake foci in bone marrow. For CT-based PD: >/= 50% decrease in SPD of up to 6 target measureable nodes and extranodal sites; non-measured lesion should be absent/normal, have regressed, but not increased; no new lesions.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax + R-CHOP 800 mg Phase II | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg + G-CHOP B
Number analyzed (Participants) | 7 | 3 | 8 | 6 | 211 | 7 | 7 | 6 | 6 | 6
Percentage of Participants | 85.71 [59.79 to 100.00] | 100.00 [100.00 to 100.00] | 87.50 [64.58 to 100.00] | 66.67 [28.95 to 100.00] | 88.99 [82.65 to 92.10] | 100.00 [100.00 to 100.00] | 75.00 [32.57 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]

19. Secondary Outcome: Percentage of Participants With CR Defined by Computed Tomography (CT) Scan Using the Modified Lugano Classification
Description: CR was defined as follows according to modified Lugano classification for CT-based response: Target nodes/nodal masses must have regressed to </= 1.5 cm in longest transverse diameter of a lesion (LDi), no extra-lymphatic sites of disease, absence of non-measured lesions, organ enlargement must have regressed to normal, no new lesions, and if the bone marrow was involved by lymphoma prior to treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
Time Frame: Baseline up to end of treatment (approx. 6 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Venetoclax + R-CHOP 800 mg Phase II
Number analyzed (Participants) | 211
Percentage of Participants | 37.4 [30.89 to 44.35]

20. Secondary Outcome: Safety: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to approximately 36 months
Population: Safety population: All patients who enrolled in the study and received any amount of venetoclax or R-CHOP/G-CHOP were included in the safety population for safety analyses
Measure: Number; unit: Percentage of Participants
Arm/Group | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax + R-CHOP 800 mg Phase II | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg + G-CHOP B
Number analyzed (Participants) | 7 | 3 | 8 | 6 | 208 | 7 | 7 | 6 | 6 | 6
Percentage of Participants | 100.00 | 100.00 | 100.00 | 100.00 | 99.0 | 100.00 | 100.00 | 100.00 | 100.00 | 100.00

21. Secondary Outcome: Safety: Percentage of Participants Maintaining Relative Dose Intensity of CHOP Chemotherapy
Description: Maintenance of relative dose intensity was defined as a dose intensity of >/= 90%.
Time Frame: Baseline up to Cycle 6 (cycle length = 21 days)
Population: Safety population: All patients who enrolled in the study and received any amount of venetoclax or R-CHOP/G-CHOP were included in the safety population for safety analyses. Overall R-CHOP and G-CHOP arms were analyzed for this outcome measure.
Measure: Number; unit: Percentage of participants
Groups:
- Venetoclax + R-CHOP Arm: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + rituximab. Each cycle consisted of 21 days.
  Phase II: Participants received 6 cycles of CHOP and 8 cycles of venetoclax (at dose determined in Phase I) + rituximab. Each cycle consisted of 21 days.
  Participants who experienced ongoing response without excessive toxicity could receive up to eight cycles of CHOP following discussion between the investigator and the Medical Monitor.
Arm/Group | Venetoclax + R-CHOP Arm | Venetoclax 600mg + G-CHOP
Number analyzed (Participants) | 232 | 32
Percentage of participants
  Cyclophosphamide: number analyzed (Participants) | 229 | 31
  Cyclophosphamide | 89.5 | 77.4
  Doxorubicin: number analyzed (Participants) | 229 | 31
  Doxorubicin | 88.6 | 77.4
  Vincristine | 86.6 | 78.1
  Prednisone: number analyzed (Participants) | 231 | 32
  Prednisone | 87.4 | 81.3

22. Secondary Outcome: Relative Dose Intensity of Venetoclax
Description: Dose intensity was categorized as < 80%, 80% to < 85%, 85% to < 90%, or >/= 90%.
Time Frame: Baseline up to Cycle 6 (cycle length = 21 days)
Population: as for outcome 20
Measure: Number; unit: Percentage of Partcipants
Groups:
- Venetoclax + G-CHOP 800mg B: Phase I: Participants received 6 cycles of CHOP and 8 cycles of venetoclax + obinutuzumab. Each cycle consisted of 21 days.
Arm/Group | Venetoclax 200 mg + R-CHOP | Venetoclax 400 mg + R-CHOP | Venetoclax 600 mg + R-CHOP | Venetoclax 800mg + R-CHOP | Venetoclax + R-CHOP 800 mg Phase II | Venetoclax 200mg + G-CHOP | Venetoclax 400mg + G-CHOP | Venetoclax 600mg + G-CHOP | Venetoclax + G-CHOP 800 mg | Venetoclax + G-CHOP 800mg B
Number analyzed (Participants) | 7 | 3 | 8 | 6 | 208 | 7 | 7 | 6 | 6 | 6
Percentage of Partcipants
  <80%: number analyzed (Participants) | 7 | 3 | 8 | 6 | 204 | 7 | 7 | 6 | 6 | 6
  <80% | 71.4 | 0.00 | 12.5 | 0.00 | 26.0 | 100.00 | 14.3 | 50.0 | 83.3 | 100.0
  80-<85%: number analyzed (Participants) | 7 | 3 | 8 | 6 | 204 | 7 | 7 | 6 | 6 | 6
  80-<85% | 0.00 | 0.00 | 12.5 | 0.00 | 3.4 | 0.00 | 14.3 | 16.7 | 0.00 | 0.00
  85-<90%: number analyzed (Participants) | 7 | 3 | 8 | 6 | 204 | 7 | 7 | 6 | 6 | 6
  85-<90% | 0.00 | 0.00 | 12.5 | 0.00 | 2.9 | 0.00 | 0.00 | 0.00 | 16.7 | 0.00
  >=90%: number analyzed (Participants) | 7 | 3 | 8 | 6 | 204 | 7 | 7 | 6 | 6 | 6
  >=90% | 28.6 | 100.00 | 62.5 | 100.00 | 67.6 | 0.00 | 71.4 | 33.3 | 0.00 | 0.00

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 67 months
Description: Safety population: All participants, who were enrolled in the study and received any amount of venetoclax or R-CHOP/G-CHOP were included in the safety population.
Arm/Group | Venetoclax 200 mg +R-CHOP | Venetoclax 400 mg +R-CHOP | Venetoclax 600 mg +R-CHOP | Venetoclax 800 mg +R-CHOP | Venetoclax 800 mg +R-CHOP Phase II | Venetoclax 200 mg +G-CHOP | Venetoclax 400 mg +G-CHOP | Venetoclax 600 mg +G-CHOP | Venetoclax 800 mg + G-CHOP A | Venetoclax 800 mg +G-CHOP B
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/3 | 1/8 | 4/6 | 33/208 | 1/7 | 1/7 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/7 | 2/3 | 4/8 | 3/6 | 116/208 | 5/7 | 4/7 | 3/6 | 5/6 | 5/6
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 8/8 | 6/6 | 204/208 | 7/7 | 7/7 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax 200 mg +R-CHOP (N=7) | Venetoclax 400 mg +R-CHOP (N=3) | Venetoclax 600 mg +R-CHOP (N=8) | Venetoclax 800 mg +R-CHOP (N=6) | Venetoclax 800 mg +R-CHOP Phase II (N=208) | Venetoclax 200 mg +G-CHOP (N=7) | Venetoclax 400 mg +G-CHOP (N=7) | Venetoclax 600 mg +G-CHOP (N=6) | Venetoclax 800 mg + G-CHOP A (N=6) | Venetoclax 800 mg +G-CHOP B (N=6)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 1 (2) | 2 (3) | 57 (89) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (3)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 19 (24) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OPTIC NEUROPATHY (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DUODENAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC DILATATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OOPHORITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SIALOADENITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADENOLYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HISTIOCYTOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CAROTID SINUS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOGLOSSAL NERVE PARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax 200 mg +R-CHOP (N=7) | Venetoclax 400 mg +R-CHOP (N=3) | Venetoclax 600 mg +R-CHOP (N=8) | Venetoclax 800 mg +R-CHOP (N=6) | Venetoclax 800 mg +R-CHOP Phase II (N=208) | Venetoclax 200 mg +G-CHOP (N=7) | Venetoclax 400 mg +G-CHOP (N=7) | Venetoclax 600 mg +G-CHOP (N=6) | Venetoclax 800 mg + G-CHOP A (N=6) | Venetoclax 800 mg +G-CHOP B (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 4 (9) | 0 (0) | 1 (1) | 2 (2) | 73 (117) | 1 (1) | 1 (1) | 1 (4) | 5 (8) | 4 (5)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 9 (10) | 0 (0) | 4 (7) | 0 (0) | 1 (1) | 0 (0)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 23 (47) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (9) | 2 (8) | 6 (18) | 3 (10) | 134 (409) | 2 (2) | 4 (17) | 5 (13) | 6 (16) | 2 (10)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (7) | 1 (2) | 3 (5) | 0 (0) | 52 (89) | 2 (3) | 3 (7) | 2 (6) | 4 (15) | 2 (5)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ICHTHYOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITREOUS FLOATERS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 14 (15) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 30 (38) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 7 (12) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 67 (78) | 6 (7) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DENTAL CYST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (10) | 2 (4) | 2 (2) | 3 (5) | 79 (133) | 5 (5) | 3 (6) | 2 (3) | 2 (4) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 22 (27) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 15 (17) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 2 (4) | 1 (1) | 5 (7) | 108 (172) | 3 (5) | 4 (7) | 3 (4) | 5 (10) | 4 (6)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 24 (29) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (6) | 64 (111) | 5 (5) | 4 (8) | 0 (0) | 4 (6) | 1 (1)
ASTHENIA (General disorders) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 33 (41) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 5 (5) | 0 (0) | 3 (3) | 2 (4) | 81 (104) | 5 (7) | 2 (2) | 2 (2) | 3 (4) | 1 (1)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 19 (28) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 23 (26) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 50 (68) | 0 (0) | 5 (7) | 2 (2) | 1 (1) | 2 (2)
UNEVALUABLE EVENT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANORECTAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 16 (18) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS ORBITAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENTEROVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ORAL FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 12 (15) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 44 (48) | 4 (4) | 1 (1) | 2 (2) | 2 (3) | 3 (4)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRACHEAL OBSTRUCTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD MAGNESIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD POTASSIUM INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINE OUTPUT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 32 (33) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 42 (45) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUID RETENTION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 35 (44) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 22 (23) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 29 (34) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 9 (10) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 12 (18) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CAROTID SINUS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 24 (33) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 19 (19) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 4 (4)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 28 (31) | 3 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2) | 1 (2) | 3 (3) | 3 (3) | 28 (33) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 18 (26) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 14 (14) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 14 (17) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
MOOD SWINGS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLADDER HYPERTROPHY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 51 (67) | 3 (3) | 2 (2) | 0 (0) | 3 (5) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 22 (24) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 11 (11) | 2 (2) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOCAL CORD DYSFUNCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 28 (29) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (9) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (15) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT02055820/Prot_002.pdf
  • Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT02055820/SAP_003.pdf